CLINICAL TRIAL: NCT02156739
Title: Radiologic Detection and Characterization of Benign and Malignant Liver Lesions in Contrast-Enhanced MRI
Brief Title: Contrast-enhanced MRI in Detecting Benign and Malignant Liver Lesions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-1157; NCI-2014-02333 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-1157 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma; Liver and Intrahepatic Bile Duct Disorder; Metastatic Malignant Neoplasm in the Liver; Primary Malignant Liver Neoplasm
MeSH Terms: conditions — Carcinoma, Hepatocellular; Digestive System Diseases | interventions — gadobutrol; gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (contrast-enhanced MRI) (Experimental): Patient receives each of these over one minute. For the gadoxetate disodium, dynamic imaging is performed immediately and imaging is performed at 20 minutes. For the gadobutrol, dynamic imaging is performed immediately.
  Interventions: Procedure: Contrast-enhanced Magnetic Resonance Imaging; Drug: Gadobutrol; Drug: Gadoxetate Disodium

INTERVENTIONS:
Procedure: Contrast-enhanced Magnetic Resonance Imaging — Undergo contrast-enhanced MRI
  Other Names: CONTRAST ENHANCED MRI; Contrast-enhanced MRI
Drug: Gadobutrol — Given IV
  Other Names: BAY86-4875; Gadavist; Gadograf; Gadovist; Protovis; ZK 135079
Drug: Gadoxetate Disodium — Given IV
  Other Names: Eovist; Gadolinium EOB DTPA; Gadolinium Ethoxybenzyl Diethylenetriaminepentaacetic Acid; Gadoxetic Acid Disodium; Gd-(S)-EOB-DTPA; Gd-EOB-DTPA; Primovist; ZK 139834

SUMMARY:
This clinical trial studies contrast-enhanced magnetic resonance imaging (MRI) in detecting nonmalignant and malignant liver lesions. Diagnostic procedures, such as MRI, may help find and diagnose nonmalignant and malignant liver lesions. Contrast agents, such as gadoxetate disodium and gadobutrol, may help doctors to see MRI images more clearly.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the specificity of contrast enhanced MRI using a liver specific agent Eovist (gadoxetate disodium) versus the combined use of Eovist and an intravascular-extracellular agent Gadavist (gadobutrol) for the radiologic detection and characterization of liver lesions via clinical stability and follow up imaging.

OUTLINE:

Patients receive gadoxetate disodium intravenously (IV) over 1 minute and undergo MRI. Patients then receive gadobutrol IV over 1 minute at the 20 minute mark during MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the most recent abdominal magnetic resonance (MR) study obtained within 3 months +/- 1 week
* Patients with renal function (estimated glomerular filtration rate [eGFR] >= 30)
* Any disease type

Exclusion Criteria:

* Pregnant women
* Patients with impaired renal function (eGFR < 30)
* Patients with surgical implants and/or metallic foreign bodies non-compatible with the MR magnet
* Patients with contraindications to the use of intravenous contrast such as allergic type reactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Specificity of combining gadoxetate disodium and gadobutrol in diagnosing tumor lesions radiologically using magnetic resonance imaging (MRI) | Up to 4 years
  Summary statistics of sensitivity, specificity, true positives, true negatives, false positives, and false negatives will be provided for gadoxetate disodium and gadoxetate disodium + gadobutrol method. Accuracy, sensitivity, specificity, positive predictive value, and negative predictive value will be estimated along with corresponding 95% confidence intervals for the two methods. Comparison between the two methods will be made following method by Obuchowski. Other statistical analyses will be carried out as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Janio Szklaruk, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org